CLINICAL TRIAL: NCT03986736
Title: Markers of Tissue Injury and Rhabdomyolysis in Patients With Major Trauma
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-11-Rhabdomyolysis; RVO-FNOs/2019-19 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2019-06-04; First posted 2019-06-14 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Tissue Injury; Major Trauma; Rhabdomyolysis
Keywords: rhabdomyolysis; tissue injury; alarmins; major trauma; acute kidney injury
MeSH Terms: conditions — Rhabdomyolysis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Two collections of full blood will be performed in the study subjects for laboratory analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with major trauma: Patients with major trauma will be included in the study.
  Interventions: Diagnostic Test: Laboratory analysis - upon admission; Diagnostic Test: Laboratory analysis - 24 hours after injury

INTERVENTIONS:
Diagnostic Test: Laboratory analysis - upon admission — Laboratory analysis will be performed upon admission of the patient to the hospital. Levels of the following parameters will be determined: HMGB-1, sCK, sMb, serum NGAL, and urine NGAL
Diagnostic Test: Laboratory analysis - 24 hours after injury — Laboratory analysis will be performed upon admission of the patient to the hospital. Levels of the following parameters will be determined: sCK, sMb, serum NGAL, and urine NGAL

SUMMARY:
Major trauma is associated with a release of alarmins (DAMPs - damage-associated molecular patterns) from the injured tissues. This process results in the activation of the immune system, which is one of the main mechanisms participating in the development of organ dysfunctions in patients with major trauma.

DETAILED DESCRIPTION:
Major trauma is associated with a release of alarmins (DAMPs - damage-associated molecular patterns) from the injured tissues. This process results in the activation of the immune system, which is one of the main mechanisms participating in the development of organ dysfunctions in patients with major trauma. Limited literary sources describe a correlation between the mitochondrial DNA (mDNA) and the value of plasma creatine kinase (sCK) (which is released from the injured muscles), which suggests a possible correlation between the number of released alarmins and the degree of rhabdomyolysis (damage of striated muscles). Rhabdomyolysis is further - due to the direct nephrotoxicity of myoglobin (sMb) released from the injured muscles - a significant factor participating in the development of acute renal failure in patients with serious injuries. Considering the fact that the serious injury need not include a vast damage of the muscle mass (especially in traumas with a minimal impairment of extremities), the correlation between the DAMPs and sCK/sMb values need not be constant in relation to the extent and localization of the injury defined with the AIS (Abbreviated Injury Scale) and ISS (Injury Severity Scale) scales. The DAMPs released from injured tissues immediately after trauma include HMGB-1 (high mobility group box 1); a correlation has been observed between the early post-injury levels of HMGB-1 and unfavorable outcome (defined with development of organ dysfunctions and increased mortality). Considering the fact that the DAMPs examination (including HMGB-1) are routinely available, and are also rather expensive, they are not a standard part of examinations performed in patients with serious trauma. Determination of correlation between HMGB-1 and the routinely available examinations of sCK and sMb would make the use of sCK and sMb examinations as direct indicators of mechanical tissue damage. Furthermore, this data has a significant descriptive impact in case of direct inclusion of sCK and sMb into predictive scoring systems, which currently do not contain relevant physiological parameters correlating with the extent of the injury.

In the second part of the study, the authors will concentrate upon evaluation of correlation of HMGB-1, serum creatine kinase and serum myoglobin in relation to the development of acute kidney injury (AKI), and in relation to the values of AKI markers, specifically NGAL (neutrophil-gelatinase associated lipocalin). The currently used AKI criteria are based upon relatively imprecise and late parameters (urine output, level of serum creatinine), and that is why AKI is identified in the clinical practice only in the stage of advanced and irreversible morphological and functional changes of kidneys.

The aims of the study are the following:

* To verify the correlation between the levels of circulating alarmins (HMGB-1) and the levels of sCK and sMb
* To identify the correlation between the levels of circulating alarmins and localization of the injury (according to AIS and ISS scoring systems)
* Mutual comparison of predictive levels of sCK and sMb in relation to the development of post-injury kidney failure
* Mutual comparison of predictive levels of sCK and sMb in relation to the serum and urine levels of AKI biomarkers
* Comparison of predictive levels of serum and urine NGAL in relation to the development of post-injury AKI

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of polytrauma
* ISS ≥ 16

Exclusion Criteria:

* history of a significant kidney impairment
* pregnancy
* injuries incompatible with life, with anticipated survival < 24 hours
* transfer to palliative care within the first 24 hours after injury
* death within the first 24 hours after injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of polytrauma.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between HMGB-1 and sCK/sMb levels | 24 hours
  Correlation between HMGB-1 and sCK/sMb levels will be assessed.
Correlation between sCK/sMb levels in relation to the degree and localisation of injury | 24 hours
  Correlation between sCK/sMb levels in relation to the degree and localisation of injury will be assessed according to the AIS and ISS scoring scales.
Mutual comparison of predictive levels of sCK/sMb in relation to post-injury acute kidney injury defined by KDIGO criteria | 8 days
  Mutual comparison of predictive levels of sCK/sMb in relation to development of post-injury acute kidney injury (defined by KDIGO criteria based both on serum creatine level investigated daily and urine output collected hourly from time of admission to Day 8 after injury) development will be assessed.
Mutual comparison of predictive levels of sCK/sMb in relation to serum and urine AKI biomarkers neutropil-gelatinase associated lipocalin (NGAL) | 8 days
  Mutual comparison of predictive levels of sCK/sMb in relation to serum and urine AKI biomarker NGAL will be assessed.
Comparison of predictive levels of serum and urine NGAL in relation to post-injury acute kidney injury development defined by KDIGO criteria. | 8 days
  Comparison of predictive levels of serum and urine NGAL in relation to post-injury acute kidney injury (defined by KDIGO criteria based both on serum creatine level investigated daily and urine output collected hourly from time of admission to Day 8 after injury) development will be assessed.

SECONDARY OUTCOMES:
Reliability of HMGB-1 in predicting major blood loss in patients with severe trauma | 8 days
  The correlation between the HMGB-1 levels and the blood loss (in ml) will be observed in patients with severe trauma
Reliability of HMGB-1 and other DAMPS in predicting organ dysfunction in intensive care unit patients | 8 days
  The correlation between HMGB-1 and other DAMPS levels and the occurrence of organ dysfunction will be observed in intensive care unit patients

CONTACTS AND LOCATIONS:
Overall Officials: Michal Frelich, MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Frelich M, Bebej M, Pavlicek J, Bursa F, Vodicka V, Svagera Z, Konde A, Jor O, Bilena M, Romanova T, Sklienka P. HMGB-1 as a predictor of major bleeding requiring activation of a massive transfusion protocol in severe trauma. Sci Rep. 2025 Feb 7;15(1):4651. doi: 10.1038/s41598-025-89139-1. PMID 39920329